CLINICAL TRIAL: NCT04891835
Title: Retrospective Analysis of naïve Patients With Age-related Macular Degeneration of the Neovascular Type and Treated With Aflibercept (Eylea®) in "Treat-and-extend" at CHU Brugmann
Brief Title: Analysis of naïve Patients With Age-related Macular Degeneration of the Neovascular Type and Treated With Aflibercept (Eylea®) in "Treat-and-extend" at CHU Brugmann
Status: Completed | Type: Observational
Sponsor: Laurence Postelmans (Other)
Responsible Party: Sponsor-Investigator, Laurence Postelmans, Head of Opthalmology clinic, Brugmann University Hospital
Organization: Brugmann University Hospital (Other)
Other Study IDs: CHUB-CHRAIBI-KAADOUD
Record Dates: First submitted 2021-05-12; First posted 2021-05-18 (Actual); Last update posted 2022-03-08 (Actual); Status verified 2022-03

CONDITIONS: Age-related Macular Degeneration
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Data extraction from medical files — Data extraction from medical files

SUMMARY:
Age-related macular degeneration (AMD) is a leading cause of blindness in people over 50. Neovascular AMD, the most serious and severe form, is characterized by the appearance, spread and growth of subretinal new vessels. One of the major molecular mediators is vascular endothelial growth factor (VEGF).

Intra-vitreous (IVI) injection of an anti-VEGF can slow the progression of neovascular AMD and stabilize vision in the majority of cases. Aflibercept (Eylea®) is one of the anti-VEGF molecules approved in Belgium to treat neovascular AMD.

At the start of its use, aflibercept was first injected monthly and then according to the PRN "reactive" protocol (Pro Renata). Over time, a new treatment strategy has emerged: the "treat-and-extend" (T&E). This is individualized patient care, the objective of which is to reduce the frequency of injections while ensuring inactivity of the disease. This begins with the loading dose, i.e. 3 injections given 4 weeks apart. Thereafter, the interval is lengthened in increments of 1 or 2 weeks provided that the visual and anatomical results remain stable. In the event of deterioration, the interval is shortened while keeping a minimum of 4 weeks between each IVI.

The efficacy and safety of aflibercept, when used in a proactive T&E regimen, was demonstrated in the randomized controlled trial, ALTAIR. However, data on T&E used in practice is still lacking. routine, and particularly the number of injections and treatment intervals over a minimum 24 month treatment period.

The aim of this retrospective study carried out at the CHU Brugmann is to determine the number of injections and the intervals necessary to have encouraging results in terms of visual acuity, over a treatment period of at least one year.

ELIGIBILITY:
Inclusion Criteria:

* Patients> 50 years old diagnosed with neovascular age related macular degeneration,
* Patients who have never received anti-VEGF treatment,
* Patients who started intra-vitreous injections of aflibercept between 01 January 2014 and November 30, 2019,
* Treatment by "treat-and-extend" directly after the loading dose of aflibercept,
* Availability of the medical file reporting treatment with aflibercept.

Exclusion Criteria:

* Participation in an interventional clinical study during treatment with aflibercept,
* Patients with ocular pathologies who required surgery during the first 24 months of treatment with aflibercept (eg advanced glaucoma or cataracts).

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients of the CHU Brugmann Hospital, > 50 years old, diagnosed with neovascular age related macular degeneration, who have never received anti-VEGF treatment, and who started intra-vitreous injections of aflibercept between 01 January 2014 and November 30, 2019.
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2021-04-13 (Actual); Primary Completion 2021-09-22 (Actual); Study Completion 2021-09-22 (Actual)

PRIMARY OUTCOMES:
Injections number (first 24 months of treatment) | first 24 months of treatment
  Number of injections during the first 24 months of treatment
Injections interval | during the 2nd year of treatment
  Last injection interval during the 2nd year of treatment, in weeks

SECONDARY OUTCOMES:
Injection number (up to 4 years of treatment) | up to 4 years of treatment
  Number of injections during the 1st, 2nd, 3rd and 4th year of treatment
Injections interval (up to 4 years of treatment) | up to 4 years of treatment
  Last injection interval during the 1st, 2nd, 3rd and 4th year of treatment (if applicable), in weeks
Most stable injection interval | up to 4 years of treatment
  Most stable injection interval during the 2nd, 3rd and 4th year of treatment (if applicable), in weeks
Overall extension interval | up to 4 years of treatment
  Expected overall extension interval: by 1 week, 2 weeks, 3 weeks or 4 weeks
Covid 19 impact | up to 4 years of treatment
  Covid19 impact on the injection interval (visits cancelled due to lock-down, shortening/increase of the injection interval due to hospital internal emergency procedures)
Number of follow-up visits | up to 4 years of treatment
  Number of follow-up visits during each year of treatment up to 4 years
Visual acuity | up to 4 years of treatment
  Visual acuity at baseline, after 90 days and at the end of each year of treatment up to 4 years
Age | Baseline
  Age of the patient at baseline
Eye lesion type | Baseline
  Eye lesion type
Fluid | up to 4 years of treatment
  Presence or absence of intra-retinal fluid, subretinal fluid, detachment of the pigment epithelium at baseline, after 90 days and at the end of each year of treatment up to 4 years
Date of first symptoms | Baseline
  Date of first symptoms of neovascular AMD
Date of first injection | Baseline
  Date of first ranibizumab injection
Retinal thickness | up to 4 years of treatment
  Retinal thickness at baseline, after 90 days and at the end of each year of treatment up to 4 years
Treatment regimen | first 12 months of treatment
  Has there been a change in treatment regimen after the first 12 months of treatment?
Number of patients stopping treatment (12-24 months) | between 12 and 24 months of treatment
  Number of patients stopping treatment between 12 and 24 months of treatment
Reason for stopping treatment (12-24 months) | between 12 and 24 months of treatment
  Reason for stopping treatment between 12 and 24 months of treatment
Number of patients stopping treatment (24-36 months) | between 24 and 36 months of treatment
  Number of patients stopping treatment between 24 and 36 months of treatment
Reason for stopping treatment (24-36 months) | between 24 and 36 months of treatment
  Reason for stopping treatment between 24 and 36 months of treatment
Number of patients stopping treatment (36-48 months) | between 36 and 48 months of treatment
  Number of patients stopping treatment between 36 and 48 months of treatment
Reason for stopping treatment (36-48 months) | between 36 and 48 months of treatment
  Reason for stopping treatment between 36 and 48 months of treatment
Number of patients stopping treatment (first 12 months) | first 12 months of treatment
  Number of patients who stopped treatment in the first 12 months
Reason for stopping treatment (first 12 months) | first 12 months of treatment
  Reason for stopping treatment in the first 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Laurence Postelmans, Study Director — CHU Brugmann
Locations (1):
- CHU Brugmann, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No